CLINICAL TRIAL: NCT00849576
Title: Effect of Treatment With Insulin VIAjectTM Compared to Regular Human Insulin and Insulin Lispro on Mealtime Blood Vessel Stress in Patients With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VIAject™-15J
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regular Human Insulin (Active Comparator): Single Injection
  Interventions: Drug: Regular Human Insulin
- Inuslin Lispro (90%) (Active Comparator): Single Injection
  Interventions: Drug: Insulin Lispro
- Insulin VIAject™ (75%) (Experimental): Single Injection
  Interventions: Drug: Insulin VIAject™ (75%)
- Insulin VIAject™ (90%) (Experimental): Single injection
  Interventions: Drug: Insulin VIAject™ (90%)

INTERVENTIONS:
Drug: Regular Human Insulin — 0.10 U/Kg- 15 minutes before ingestion of a standardized liquid meal.
  Arms: Regular Human Insulin
Drug: Insulin Lispro — 90% of Regular Human Insulin dose administer immediately before ingestion of a standardized liquid meal.
  Arms: Inuslin Lispro (90%)
Drug: Insulin VIAject™ (75%) — 75 % of Regular Human Insulin dose administer immediately before ingestion of a standardized liquid meal
  Arms: Insulin VIAject™ (75%)
Drug: Insulin VIAject™ (90%) — 90 % of Regular Human Insulin dose administer immediately before ingestion of a standardized liquid meal
  Arms: Insulin VIAject™ (90%)

SUMMARY:
The purpose of this study is to compare the effects of insulin VIAject with Regular Human Insulin and Insulin Lispro on measures of mealtime blood vessel stress and blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus according to the ADA criteria
2. HbA1c between 6.5 % and 9.9 %
3. Treatment with sulfonylurea and/or metformin in a stable dosage within the last 3 months
4. Age between 40 and 75 years
5. BMI < 40

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Pre-treatment with insulin within the last 6 months prior to screening
3. Pre-treatment with PPARy-agonists or glucosidase inhibitors within the last 4 weeks prior to screening
4. Untreated hypertension stage II-III according to WHO criteria
5. Planned or anticipated change in antidiabetic and/or concomitant medication during study participation
6. Total cholesterol > 300 mg/dl (anamnestically)
7. Major micro- or macrovascular complications as judged by the investigator
8. Tobacco use within the last 6 months prior to screening
9. Drugs with major impact on endothelial function like nitrates etc.
10. History of drug or alcohol abuse which in the opinion of the investigator will impair subject safety or protocol compliance
11. History of hypersensitivity to the study drugs or to drugs with similar chemical structures
12. History of severe or multiple allergies
13. Treatment with any other investigational drug within 3 months prior to screening
14. Progressive fatal disease
15. History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.1 mg/dL in women and > 1.5 mg/dL in men), neurological, psychiatric and/or haematological disease as judged by the investigator
16. Pregnancy or breast feeding
17. Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomised partner
18. Lack of compliance or other similar reason that at the discretion of the investigator precludes satisfactory participation in the study
19. Hypopotassemia (K<3.5 mmol /l)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Postprandial time course of Asymmetric dimethyl arginine (ADMA) after injection of insulin VIAjectTM compared with regular human insulin and insulin lispro. | 0 - 240 minutes

SECONDARY OUTCOMES:
The secondary objectives are to evaluate the postprandial time course of arterial elasticity (pulse wave analysis; PWA), blood glucose, insulin, intact proinsulin, nitrotyrosine, glucagon, ICAM-1, VCAM, E-selectin. | 0 - 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, MD, Principal Investigator — IKFE Institute for Clinical Research and Development
Locations (1):
- IKFE, Parcusstrasse 8, Mainz, Germany